CLINICAL TRIAL: NCT01588821
Title: Phase II Trial of Cabozantinib (XL184) in Patients With Advanced Solid (Non-breast, Non-prostate) Malignancies and Bony Metastases
Brief Title: Cabozantinib in Advanced Solid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rebecca Suk Heist, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-091
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Lung Cancer; Solid Tumor (Not Breast or Prostate Cancers)
Keywords: Metastatic; Refractory; Relapsed
MeSH Terms: conditions — Lung Neoplasms; Prostatic Neoplasms; Neoplasm Metastasis; Recurrence | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Cabozantinib
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — 60 mg daily by mouth
  Other Names: XL184

SUMMARY:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if the drug is effective for treating different types of cancer. It also means that the FDA has not approved the drug for this type of cancer, or for any use outside of research studies.

When cancer spreads from the primary tumor, one of the most commons sites it spreads to is bone. When cancer spreads to bone there can be significant symptoms such as pain.

Cabozantinib works by blocking signaling that leads to cancer growth as well as blocking the growth of new blood vessels (angiogenesis) that help to feed a tumor. Cabozantinib has been studied or is being studied in research studies as a possible treatment for various types of cancer, including prostate cancer, brain cancer, thyroid cancer, lung cancer and kidney cancer.

Previous clinical research studies indicate that cabozantinib may also have activity against cancer once it has spread to the bones.

The purpose of this study is to find out if cabozantinib is effective in treating cancer that has spread to the bone.

DETAILED DESCRIPTION:
Cabozantinib is a tablet that the subject will take by mouth. The subject will take it once per day. The study treatment with cabozantinib will be divided into 28 day cycles. A member of the study staff will give the subject a drug diary and explain to the subject how to use it to record doses of cabozantinib. This diary will also contain specific instructions about how the subject take cabozantinib.

Every 28 days the subject will undergo the following procedures: Physical examination, questions about any side effects the subject may have, blood samples for routine laboratory tests and research tests, urine sample, electrocardiogram (EKG), and questionnaires to measure quality of life and level of pain. Every two months the subject will undergo a CT scan or MRI to evaluate the subjects disease.

The investigators would like the subject to return to the study clinic for follow-up procedures about 4-5 weeks after the last dose of cabozantinib.

The subject can continue to receive the study drug for as long as their disease does not worsen and the subject do not experience unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of a solid tumor (not breast or prostate) that is metastatic and refractory to or progressed following standard therapies
* Has bony metastases
* Agree to use medically accepted methods of contraception

Exclusion Criteria:

* Pregnant or breastfeeding
* Received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents within 3 weeks of study entry(6 weeks for nitrosoureas/mitomycin C)
* Received radiation to the thoracic cavity/GI tract (within 3 months of study entry), to bone or brain metastasis (within 14 days) or to any other site within 28 days
* Received prior treatment with small molecule kinase inhibitor or hormonal therapy within 14 days/5 half-lives
* Received therapy with another investigational agent within past 28 days
* Has not recovered from toxicities due to prior therapies
* Primary brain tumor
* Active brain metastases or epidural disease
* Uncontrolled significant intercurrent or recent illness
* Allergy or hypersensitivity to components of the study treatment formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-06; Primary Completion 2017-01 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Heist, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabozantinib
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib
Number analyzed (Participants) | 37
Age, Continuous [Mean (Full Range); unit: years] | 54.4 [18 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 37
Diagnosis [Count of Participants; unit: Participants]
  Sarcoma | 14
  Renal Cell Carcinoma | 7
  Non-Small cell lung cancer | 5
  Head and neck carcinoma | 4
  Thyroid Cancer | 2
  Melanoma | 2
  Adenoid Cystic Carcinoma | 1
  Metastatic chondroblastoma | 1
  Chordoma | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bone Bio-marker Response
Description: Effect of cabozantinib on bone biomarkers of osteoblast and osteoclast activity. The bio-markers of interest were serum C-terminal telopeptide (Ctx), urine N-terminal telopeptide (Ntx), serum (Ntx). Participants were considered to have a response if there was at least a 40% decrease in the bio-marker concentration.
Time Frame: 8 Weeks
Population: Only 19 participants were evaluable for determination of response by bone bio-markers
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 19
Participants
  Serum Ctx | 13
  Urine Ntx | 9
  Serum Ntx | 8

2. Secondary Outcome: Number of Patients With Skeletal-related Events (SRE)
Description: The number of patients that experience a SRE in patients treated with cabozantinib (SRE defined as pathologic fracture, cord compression, radiation or surgery to bone, hypercalcemia)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 37
Participants | 0

3. Secondary Outcome: Quality of Life as Assessed by FACT-G
Description: Quality of life as measured by the Functional Assessment of Cancer Therapy - General (FACT-G). FACT-G assesses patients' physical, social/family, emotional, and functional well-being. The total score can range from 0 to 108, with lower scores indicating higher quality of life. Patients without QOL scores at cycle 3 day 1 had their score from their last assessment carried forward.
Time Frame: From baseline to Cycle 3 Day 1 (approximately 2 months)
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Cabozantinib
Number analyzed (Participants) | 37
units on a scale
  Baseline | 56 [41 to 63]
  Cycle 3 Day 1 | 56 [20 to 71]

4. Secondary Outcome: Overall Tumor Response Rate
Description: The number of participants with a complete or partial response as measured by bone scan or PET-CT scan using. Response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
  * Complete Response (CR): Disappearance of all target lesions
  * Partial Response (PR): At least a 30% decrease in the sum of the Longest Diameter (LD) of target lesions, taking as reference the baseline sum LD
Time Frame: 2 years
Population: The 20 participants that were able to be evaluated for response. The other 17 participants had bone only disease
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 20
Participants
  Complete Response | 0
  Partial Response | 3

5. Secondary Outcome: MET Amplification in Tumor Sample
Description: Response will be correlated with specific tumor genotype (MET amplification).
Time Frame: 2 years
Population: MET amplification testing was not done due to insufficient tumor material available for testing
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Response to Cabozantinib in Bone Metastatic Disease
Description: Response to cabozantinib in bone metastatic disease as measured by bone scan or PET-CT scan
Time Frame: 2 years
Population: Bone scan response assessment not done
Arm/Group | Cabozantinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to SRE
Description: Time to SRE in patients treated with cabozantinib (SRE defined as pathologic fracture, cord compression, radiation or surgery to bone, hypercalcemia)
Time Frame: 2 years
Population: No SRE events occurred
Arm/Group | Cabozantinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Beginning at the start of treatment, adverse events are assessed every 2 weeks for the first 3 months and then on a monthly basis up until 30 days after the last dose of Cabozantinib is received. Overall adverse event data collection is ongoing. Data represents all adverse events collected at the time of initial data analysis.
Description: Participants are assessed with the use of physical exams, laboratory tests, electrocardiograms (EKG), and by participant self reporting.
Arm/Group | Cabozantinib
All-Cause Mortality (participants affected / at risk) | 4/37
Serious Adverse Events (participants affected / at risk) | 9/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (N=37)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (N=37)
Anemia (Blood and lymphatic system disorders) | 8 (10)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3 (3)
Cardiac disorders - Other, specify (Cardiac disorders) | 5 (5)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 24 (42)
Fever (General disorders) | 3 (4)
Flu like symptoms (General disorders) | 2 (2)
Malaise (General disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 4 (5)
Pain (General disorders) | 17 (21)
General disorders and administration site conditions - Other, (General disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 13 (18)
Hypothyroidism (Endocrine disorders) | 11 (11)
Endocrine disorders - Other, specify (Endocrine disorders) | 2 (2)
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 21 (22)
Diarrhea (Gastrointestinal disorders) | 18 (27)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 12 (16)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 17 (23)
Oral dysesthesia (Gastrointestinal disorders) | 3 (4)
Oral pain (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 7 (7)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 4 (4)
Meningitis (Infections and infestations) | 2 (2)
Prostate infection (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 5 (5)
Urinary tract infection (Infections and infestations) | 3 (4)
Infections and infestations - Other, specify (Infections and infestations) | 5 (5)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 13 (15)
Alkaline phosphatase increased (Investigations) | 10 (11)
Aspartate aminotransferase increased (Investigations) | 19 (22)
CPK increased (Investigations) | 3 (3)
Lipase increased (Investigations) | 5 (8)
Platelet count decreased (Investigations) | 5 (8)
Serum amylase increased (Investigations) | 3 (5)
Weight loss (Investigations) | 10 (14)
White blood cell decreased (Investigations) | 3 (3)
Investigations - Other, specify (Investigations) | 7 (8)
Anorexia (Metabolism and nutrition disorders) | 12 (17)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (18)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 6 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (17)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Musculoskeletal and connective tissue disorder - (Musculoskeletal and connective tissue disorders) | 7 (9)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 5 (6)
Glaucoma (Eye disorders) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 5 (5)
Depression (Psychiatric disorders) | 9 (9)
Insomnia (Psychiatric disorders) | 12 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 6 (6)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 13 (13)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2)
Hypertension (Vascular disorders) | 23 (32)
Hypotension (Vascular disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes